CLINICAL TRIAL: NCT04384757
Title: Comparison of Laparoscopic Versus Open Distal Gastrectomy for T4a Gastric Cancer: a Prospective Randomized Control Trial
Brief Title: Comparison of Open and Laparoscopic Distal Gastrectomy for T4a Gastric Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Responsible Party: Principal Investigator, VoDuy Long, Deputy Head of GI Surgery Department, University Medical Center Ho Chi Minh City (UMC)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMC-UPPERGI-01
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; laparoscopic gastrectomy; T4a stage
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gastroenterostomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open distal gastrectomy (Active Comparator): An incision of 15~20 cm length is made in the abdominal midline . Standard distal gastrectomy and omentectomy will be performed with D2 lymph node dissection (around common hepatic artery, celiac artery, proximal part of splenic artery, proper hepatic artery) . As a general rule, Billroth II method was used for gastric reconstruction for most cases
  Interventions: Procedure: Distal gastrectomy
- Laparoscopic distal gastrectomy (Experimental): 5 trocar were used. The gastrocolic ligament was divided along the border of the transverse colon. ligating the left gastroepiploic vessels to remove group 4sb.
  The right gastroepiploic vein was divided and the right gastroepiploic and the inferior pyloric artery were vascularized and cut at their origin from the gastroduodenal artery, just above the pancreatic head, to dissect group 6.
  The dissection was continued along the hepatoduodenal ligament to removed group 5 and group 12a and along the common hepatic artery to remove group 8a and along the celiac axis to remove group 9.
  The left gastric vein was prepared and separately divided and then the left gastric artery was vascularized to remove group 7.
  The dissection was continued upward along the proximal branches of splenic vessels to remove group 11p and along the lesser curvature to remove group 1,3.
  As a general rule, Billroth II method was used for gastric reconstruction for most cases
  Interventions: Procedure: Distal gastrectomy

INTERVENTIONS:
Procedure: Distal gastrectomy — Distal gastrectomy and standard D2 lymphadenectomy

SUMMARY:
There are more than 75% of patients with gastric cancer who are diagnosed in advanced stage in Vietnam, most of cases in T4a. The purpose of this study is to compare the technical feasibility, early and long term outcomes of open and laparoscopic distal gastrectomy for gastric adenocarcinoma in T4A stage

DETAILED DESCRIPTION:
Gastric cancer poses a significant public health problem. It is one of the most common cancers in Vietnam . Despite recent advances in multimodality treatment and targeted therapy, surgery remains the first option of treament for this disease. For resectable gastric cancer, complete removal of macroscopic and microscopic lesions and/or combined resections and also regional or extended lymphadenectomy should represent in the world now. Since laparoscopic gastrectomy for early gastric cancer (EGC) was firstly reported in 1994 , this technique has become standard for treatment of EGC due to the many advantages of mininally invasive surgery and also in oncologic outcomes.

Laparoscopic gastrectomy for advanced gastric cancer AGC was first applied by Uyama in 2000, and then, many surgeons have used it for treatment of AGC, especially in Japan, Korea and China. However, the real role of laparoscop for treament of (AGC) is still controversial in term of technical feasibility, safety and oncologic aspect.

Paragastric inflammatory strands may occur in T4a tumor so that laparoscopic technique is difficult to radically perform. Peritoneal seeding of malignant cells, intra- and postoperative complications, trocarts metastasis may risk during procedures. Despite, some studies have demonstrated the safety and the short-term benefits of LG for T4a gastric cancer, the number of these studies and sample sizes have been still inadequate to give good evidence for applying it. and long-term oncologic outcomes

There are more than 75% of patients with gastric cancer who are diagnosed in advanced stage in Vietnam, most of cases in T4a. The purpose of this study is to compare the technical feasibility, early and long term outcomes of open and laparoscopic distal gastrectomy for gastric adenocarcinoma in T4A stage.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic finding by gastric endoscopy: confirmed gastric adenocarcinoma
* Age: 18 - 80 year old
* Tumor located at the middle or lower third of the stomach
* Preoperative cancer stage (CT scan stage): cT4aN0M0, cT4aN1M0, cT4aN2M0, cT4aN3M0
* ASA score: ≤ 3
* Informed consent patients (explanation about our clinical trials is provided to the patients or patrons, if patient is not available)

Exclusion Criteria:

* Concurrent cancer or patient who was treated due to other cancer before the patient was diagnosed gastric cancer
* Had another treatment methods, such as chemotherapy, immunotherapy, or radiotherapy
* Pregnant patient
* Combined resection
* Total gastrectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
3 year overall survival by Kaplan Mayer | 3 year after surgery
  The percentage of people in this study who are alive three years after surgery.
3 year relapse-free survival by Kaplan Mayer | 3 year after surgery
  The percentage of people in this study who are alive without recurrence three years after surgery.

SECONDARY OUTCOMES:
operative morbidity | 30 days after surgery
  The rate of postoperative bleeding and the rate of postoperative leakage
operative mortality | 30 days after surgery
  The rate of postoperative dead
hospital stay | 30 days after surgery
  The number of days between surgery and discharge
operative time | intraoperative
  The duration of a surgical procedure in minutes.
Resected lymph nodes | intraoperative
  the number of lymph nodes harvested after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Long D. Vo, PhD, MD, Principal Investigator — University Medical Center, 215 Hong Bang street, Dist. 5, HCM city, VN
Locations (1):
- University Medical Center, Ho Chi Minh City, Ho Chi Minh, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided
Waiting for the results of this study

REFERENCES:
- [Derived] Dat TQ, Thong DQ, Nguyen DT, Hai NV, Phuoc TD, Anh NVT, Bac NH, Long VD. Laparoscopic vs Open Distal Gastrectomy With D2 Lymphadenectomy for Clinical T4a Gastric Cancer: The UMC-UPPERGI-01 Randomized Clinical Trial. JAMA Surg. 2026 Jan 1;161(1):9-18. doi: 10.1001/jamasurg.2025.4929. PMID 41222957
- [Derived] Dat TQ, Thong DQ, Nguyen DT, Hai NV, Vuong NL, Bac NH, Long VD. Laparoscopic versus open distal gastrectomy with d2 lymphadenectomy in treatment of locally T4A gastric cancer: the protocol of a randomized controlled trial. BMC Surg. 2025 May 2;25(1):193. doi: 10.1186/s12893-025-02933-6. PMID 40316937